CLINICAL TRIAL: NCT00508118
Title: NICardipine Neuroprotection in AortiC Surgery (NICNACS)
Acronym: NICNACS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: 3/7 subjects experienced hypotension. Study was terminated.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00001612
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2013-01

CONDITIONS: Aortic Aneurysm, Thoracic
Keywords: Aortic Arch Reconstruction Surgery
MeSH Terms: conditions — Aortic Aneurysm, Thoracic | interventions — Nicardipine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Nicardipine
  Interventions: Drug: Nicardipine
- 2 (Placebo Comparator): 0.9% saline
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Nicardipine — on bypass
  Arms: 1
Drug: 0.9% saline — on bypass
  Arms: 2

SUMMARY:
Objective

The objective of this study is to discover whether an infusion of nicardipine is able to reduce the time taken to achieve electrocerebral silence (ECS) during cardiopulmonary bypass (CPB) for aortic surgery.

Hypothesis

By inhibiting cold-induced cerebral vasoconstriction, nicardipine will maintain cerebral blood flow and allow more rapid cooling of the brain during CPB. This will manifest as a reduction in the time taken to achieve ECS and also as a reduction in overall CPB time.

DETAILED DESCRIPTION:
Patients undergoing thoracic aortic surgery at Duke University Medical Center (DUMC) requiring hypothermic circulatory arrest (HCA) and neurophysiologic monitoring (NIOM) will give written informed consent and be enrolled into the study. Exclusion criteria will include previously documented allergy to nicardipine and age less than 18 years. Patients will then be randomized to one of two study groups: general anesthesia with or without nicardipine. Pre-operatively they will undergo clinical evaluation determined by the attending surgeon and anesthesiologist. During the pre-induction time period, all usual monitors and intravenous devices will be placed at the discretion of the attending anesthesiologist. In addition to the standard anesthetic monitors (Bispectral Index [BIS] and cerebral oximetry), transcranial Doppler (TCD) will be placed. Furthermore, the neurophysiology technician will place both standard EEG and somatosensory evoked potential (SSEP) electrode configurations. During the pre-induction time period, midazolam use will be at the discretion of the anesthesiologist but will be limited to a maximum dose of 0.1 mg/kg; other benzodiazepines will not be allowed. Opioid (fentanyl) administration will be at the discretion of the anesthesiologist. Total benzodiazepine and opioid doses will be recorded and converted to midazolam and fentanyl equivalents for subsequent analysis.

When ready, patients will be transported into the operating room and anesthesia will be induced. Induction will consist of propofol (1 - 5 mg/kg single intravenous bolus), fentanyl and vecuronium for neuromuscular blockade. Other drugs and dosages of opioids and neuromuscular blockers are at the discretion of the anesthesiologist. After induction and tracheal intubation, patients will receive maintenance anesthesia of 0.5 minimal alveolar concentration (MAC) isoflurane in a 50% air/oxygen balanced mixture supplemented with fentanyl at the discretion of the anesthesiologist. At the onset of cardiopulmonary bypass (CPB), study drug (nicardipine or equivalent volume of placebo - 0.9% saline) infusion at 5 mg/hr will be initiated, and patients will receive 0.5 MAC isoflurane in the CPB circuit sweep gas. Bolus doses of 100mcg phenylephrine will be administered to both groups in order to maintain a constant mean arterial pressure of at least 50 mmHg. Cooling will occur primarily through the CPB machine. When the patient's brain temperature reaches 28o C, isoflurane (via the pump) will be reduced to 0.25 MAC. When ECS on EEG and ablation of cortical responses on SSEP have both occurred, CPB and study drug infusion will be halted, and thoracic aortic surgery will be commenced. After aortic repair has occurred, CPB and study drug infusion at 5 mg/hr will be reinstated, anesthesia administration resumed, and the patient actively rewarmed. When the patient's brain temperature reaches 28o C (as recorded by nasopharyngeal temperature), patients will receive 0.5 MAC isoflurane. After the patient has been fully re-warmed and is ready for separation from CPB, study drug infusion will be halted. At this point, but not before, commercially available nicardipine may be infused if so desired. 10 ml blood samples will be drawn from the pump at baseline and 15 minute intervals thereafter until HCA is achieved. When the pump is restarted, further samples will be drawn at 15 minute intervals until the patient separates from CPB after which no further samples will be taken. One sample of 10 ml will be drawn from the retrograde cardioplegia line immediately after placement (baseline) and one sample will be drawn immediately prior to separation from CPB. In total, approximately 100 ml of blood will be drawn from the patient for research purposes. This volume represents a tiny percentage of the excess volume associated with the pump prime, and is insignificant in terms of its effect on hemodynamics.

Baseline patient characteristics will be collected in the pre-operative period and will include age, sex, weight, height, blood pressure, heart rate, temperature, comorbidities, type of aortic disease, and American Society of Anesthesiologists (ASA) grade. Prior to initiation of CPB, several factors will be recorded including arterial blood pressure, heart rate, cerebral oximetry, bispectral index score (BIS), latency & amplitude of SSEP, frequency of EEG background, cerebral blood flow assessed by middle cerebral artery (MCA) velocity on TCD, and nasopharyngeal temperature. During cooling, BIS scores, cerebral oximetry, and MCA velocity by TCD will be noted for each 0.5o C decrement in nasopharyngeal temperature; the duration from CPB initiation to 3 characteristic EEG changes (1. rhythmic delta, 2. Generalized periodic epileptiform discharge (GPED), 3. burst suppression) as defined by the neurophysiologist, the duration from CPB initiation to 2 characteristic SSEP changes (1. latency increase of >10%, 2. amplitude decrease of 50% from baseline), and hemodynamics at each 1o C nasopharyngeal temperature drop will also be recorded. At the time of HCA, several factors will be documented including nasopharyngeal temperature, duration from CPB initiation (the primary endpoint measure), total opioid doses, cerebral oximetry, BIS score, MCA velocity by TCD, hemodynamics. During rewarming, factors will be documented in the same fashion and at the same intervals as during cooling. At the first attempt at separation from CPB, documented factors will include BIS score, cerebral oximetry, MCA velocity by TCD, duration from CPB reinstitution to first attempt at separation, total dose of study drug, nasopharyngeal temperature, and hemodynamics. Finally, in addition to any Adverse Events (AEs) that may have occurred, data relating to length of ICU stay, length of hospital stay, in-hospital mortality, in-hospital acute kidney injury (defined as a 50% rise from baseline in serum creatinine, and of at least 0.3 mg/dl or need for dialysis), in-hospital stroke, in-hospital myocardial infarction, and discharge disposition from hospital (home, skilled nursing facility, other institution) will be recorded postoperatively.

With the exception of the on-pump blood draws, in this protocol there are no additional procedures or safety measures indicated or necessary for the purpose of research only. All anesthetic regimens and monitoring techniques are currently standard of care. Nicardipine infusion is currently widely used during cardiac anesthesia and post-operative cardiac recovery.

ELIGIBILITY:
Inclusion Criteria:

* All adult (>18 years) patients at Duke University Medical Center (DUMC) presenting for elective aortic surgery scheduled to include a period of deep hypothermic circulatory arrest.

Exclusion Criteria:

* Failure to provide written informed consent
* Emergency operation
* Documented allergy to nicardipine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andy Shaw, M. D., Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Guerit JM, Verhelst R, Rubay J, el Khoury G, Noirhomme P, Baele P, Dion R. The use of somatosensory evoked potentials to determine the optimal degree of hypothermia during circulatory arrest. J Card Surg. 1994 Sep;9(5):596-603. doi: 10.1111/j.1540-8191.1994.tb00892.x. PMID 7994101
- [Background] Ghariani S, Liard L, Spaey J, Noirhomme PH, El Khoury GA, de Tourtchaninoff M, Dion RA, Guerit JM. Retrospective study of somatosensory evoked potential monitoring in deep hypothermic circulatory arrest. Ann Thorac Surg. 1999 Jun;67(6):1915-8; discussion 1919-21. doi: 10.1016/s0003-4975(99)00413-0. PMID 10391338
- [Background] Fleck TM, Czerny M, Hutschala D, Koinig H, Wolner E, Grabenwoger M. The incidence of transient neurologic dysfunction after ascending aortic replacement with circulatory arrest. Ann Thorac Surg. 2003 Oct;76(4):1198-202. doi: 10.1016/s0003-4975(03)00832-4. PMID 14530011
- [Background] Dahlbacka S, Makela J, Kaakinen T, Alaoja H, Heikkinen J, Laurila P, Kiviluoma K, Salomaki T, Tuominen H, Ohtonen P, Lepola P, Biancari F, Juvonen T. Propofol is associated with impaired brain metabolism during hypothermic circulatory arrest: an experimental microdialysis study. Heart Surg Forum. 2006;9(4):E710-8; discussion E718. doi: 10.1532/HSF98.20061022. PMID 16844626
- [Background] Hirotani T, Kameda T, Kumamoto T, Shirota S. Aortic arch repair using hypothermic circulatory arrest technique associated with pharmacological brain protection. Eur J Cardiothorac Surg. 2000 Nov;18(5):545-9. doi: 10.1016/s1010-7940(00)00533-9. PMID 11053815
- [Background] Khaladj N, Peterss S, Oetjen P, von Wasielewski R, Hauschild G, Karck M, Haverich A, Hagl C. Hypothermic circulatory arrest with moderate, deep or profound hypothermic selective antegrade cerebral perfusion: which temperature provides best brain protection? Eur J Cardiothorac Surg. 2006 Sep;30(3):492-8. doi: 10.1016/j.ejcts.2006.05.031. Epub 2006 Jul 20. PMID 16857368
- [Background] Levy WJ, Pantin E, Mehta S, McGarvey M. Hypothermia and the approximate entropy of the electroencephalogram. Anesthesiology. 2003 Jan;98(1):53-7. doi: 10.1097/00000542-200301000-00012. PMID 12502979
- [Background] Pokela M, Jantti V, Lepola P, Romsi P, Rimpilainen J, Kiviluoma K, Salomaki T, Vainionpaa V, Biancari F, Hirvonen J, Kaakinen T, Juvonen T. EEG burst recovery is predictive of brain injury after experimental hypothermic circulatory arrest. Scand Cardiovasc J. 2003 Jun;37(3):154-7. doi: 10.1080/14017430310006956. PMID 12881157
- [Background] Puri GD, Bagchi A, Anandamurthy B, Dhaliwal RS. The Bispectral Index and induced hypothermia--electrocerebral silence at an unusually high temperature. Anaesth Intensive Care. 2003 Oct;31(5):578-80. doi: 10.1177/0310057X0303100515. PMID 14601285
- [Background] Sakamoto T, Hatsuoka S, Stock UA, Duebener LF, Lidov HG, Holmes GL, Sperling JS, Munakata M, Laussen PC, Jonas RA. Prediction of safe duration of hypothermic circulatory arrest by near-infrared spectroscopy. J Thorac Cardiovasc Surg. 2001 Aug;122(2):339-50. doi: 10.1067/mtc.2001.115242. PMID 11479508
- [Background] Speziali G, Russo P, Davis DA, Wagerle LC. Hypothermia enhances contractility in cerebral arteries of newborn lambs. J Surg Res. 1994 Jul;57(1):80-4. doi: 10.1006/jsre.1994.1114. PMID 8041154
- [Background] Stecker MM, Cheung AT, Pochettino A, Kent GP, Patterson T, Weiss SJ, Bavaria JE. Deep hypothermic circulatory arrest: I. Effects of cooling on electroencephalogram and evoked potentials. Ann Thorac Surg. 2001 Jan;71(1):14-21. doi: 10.1016/s0003-4975(00)01592-7. PMID 11216734
- [Background] Stecker MM, Cheung AT, Pochettino A, Kent GP, Patterson T, Weiss SJ, Bavaria JE. Deep hypothermic circulatory arrest: II. Changes in electroencephalogram and evoked potentials during rewarming. Ann Thorac Surg. 2001 Jan;71(1):22-8. doi: 10.1016/s0003-4975(00)02021-x. PMID 11216751
- [Background] Stecker MM, Escherich A, Patterson T, Bavaria JE, Cheung AT. Effects of acute hypoxemia/ischemia on EEG and evoked responses at normothermia and hypothermia in humans. Med Sci Monit. 2002 Apr;8(4):CR223-8. PMID 11951061

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicardipine: Nicardipine infusion before bypass
  After enrollment of 7 patients the operating surgeon (also a study collaborator) commented that 3 of the patients appeared to have required more vasopressor support than was usual in his practice and so these patient allocations were unblinded. All 3 had been randomized to receive nicardipine. Thus, even if all 7 enrolled so far had been randomized to active drug this would have meant an incidence of at least 37.5% requiring increased vasopressor use. After discussion with the surgeon (Dr Hughes), and the other co-investigators it is the decision of the study team and PI that this protocol is not able to safely answer the research question posed and thus further enrollment would be inappropriate. One subject cannot be accounted for as to treatment arm. No further documentation available.
- 0.9% Saline: 0.9% saline (placebo) infusion before bypass
Period: Overall Study
Arm/Group | Nicardipine | 0.9% Saline
Started | 3 | 4 (Documentation is not available for the 7th subject and treatment arm.)
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nicardipine: Nicardipine infusion before bypass
- 0.9% Saline: 0.9% saline (placebo) before bypass
- Total: Total of all reporting groups
Arm/Group | Nicardipine | 0.9% Saline | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 3 |  | 3
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (5) |  | 50 (5)
Gender [Number; unit: participants]
  Female | 1 |  | 1
  Male | 2 |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Duration From Initiation of Cardiopulmonary Bypass (CPB) to Electrocerebral Silence (ECS), Defined as no Discernable Electroencephalographic Activity at an Amplification of 2 Micro Volts (μV)/mm, Confirmed for 3 Minutes
Time Frame: Day of surgery
Population: 3 SUBJECTS PER PROTOCOL.
Measure: Median (95% Confidence Interval); unit: Time (minutes)
Groups:
- NICARDIPINE GROUP: Nicardipine prior to bypass
Arm/Group | NICARDIPINE GROUP
Number analyzed (Participants) | 3
Time (minutes) | 45 [35 to 56]

2. Secondary Outcome: Temperature at Which ECS Occurs
Time Frame: Day of surgery through discharge
Population: No participants analyzed due to study terminated early.
Arm/Group | Nicardipine | 0.9% Saline
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Temperature at Which Ablation of(SSEP)Occurs
Time Frame: Day of surgery through discharge
Population: No participants were analyzed due to study terminated early.
Arm/Group | Nicardipine | 0.9% Saline
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time Points of EEG Patterns
Time Frame: Day of surgery through discharge
Population: No participants were analyzed due to study terminated early.
Arm/Group | Nicardipine | 0.9% Saline
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time Points for SSEP Latency and Amplitude Changes
Time Frame: Day of surgery through discharge
Population: No participants were analyzed due to study terminated early.
Arm/Group | Nicardipine | 0.9% Saline
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Bispectral Index Scores (BIS)
Time Frame: Day of surgery through discharge
Population: No participants were analyzed due to study terminated early.
Arm/Group | Nicardipine | 0.9% Saline
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Cerebral Oximetry Measurements
Time Frame: Day of surgery through discharge
Population: No participants were analyzed due to study terminated early.
Arm/Group | Nicardipine | 0.9% Saline
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Transcranial Doppler Measurements
Time Frame: Day of surgery through discharge
Population: No participants were analyzed due to study terminated early.
Arm/Group | Nicardipine | 0.9% Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Nicardipine | 0.9% Saline
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicardipine (N=3) | 0.9% Saline (N=3)
Hypotension (Cardiac disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early because of safety concerns in the active treatment group. In 3 patients randomized, the blind was broken in 3 because of refractory hypotension and acidosis requiring vasopressor therapy. All 3 were on active drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No